CLINICAL TRIAL: NCT01728311
Title: An Open-label Phase I Dose-escalation Study to Characterize the Safety, Tolerability, Pharmacokinetics, and Maximum Tolerated Dose of BAY 1082439 Given Once Daily Continuously or in an Intermittent Dosing Schedule in Subjects With Advanced Malignancies
Brief Title: Open Label Study of BAY1082439 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15734
Record Dates: First submitted 2012-11-07; First posted 2012-11-19 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: BAY1082439

INTERVENTIONS:
Drug: BAY1082439 — BAY1082439 will be given orally once daily with a 21 days cycle. Dose will be started from 15mg.

SUMMARY:
The purpose of this study is to determine the safety, tolerability and the pharmacokinetics of BAY1082439

ELIGIBILITY:
Inclusion Criteria:

* Subjects with advanced, histologically or cytologically confirmed solid tumors, refractory to any standard therapy, have no standard therapy available, or subjects must have actively refused any treatment which would be regarded standard, and / or if in the judgment of the investigator, experimental treatment is clinically and ethically acceptable

  * Expansion phase only: Subjects with histologically or cytologically confirmed, locally advanced or metastatic endometrial cancer or breast cancer or iNHL, who are refractory to or have exhausted all available therapies
* International normalized ratio (INR) and partial thromboplastin time (PTT) <1.5 x ULN [Subjects on anticoagulation with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.] For subjects on warfarin, close monitoring of at least weekly evaluations will be performed until INR is stable based on a measurement at pre-dose, as defined by the local standard of care
* Measurable or evaluable disease
* Life expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* History of cardiac disease: congestive heart failure > New York Heart Association (NYHA) Class II, unstable angina (anginal symptoms at rest), new-onset angina (within the past 3 months prior to the first dose of study drug), myocardial infarction within the past 6 months prior to the first dose of study drug, or cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management
* History of diabetes mellitus or gestational diabetes mellitus
* Fasting blood glucose level >125 mg/dL or HbA1c 7% at screening
* Active clinically serious infections > Grade 2
* History of organ allograft
* Seizure disorder requiring therapy (such as steroids or anti-epileptics)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11-21 (Actual); Primary Completion 2016-06-03 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to 2 years
Maximum tolerated dose of BAY1082439 | Up to 1 year
Maximum observed plasma concentration (Cmax) of BAY1082439 after a single dose | Serial PK samples will be selected during cycle 1 day 1 (pre-dose and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose) and sparse samples during the rest of the cycle as well as in cycle 2
Time to Cmax (tmax) of BAY1082439 after a single dose | Serial PK samples will be selected during cycle 1 day 1 (pre-dose and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose) and sparse samples during the rest of the cycle as well as in cycle 2
Area under the plasma concentration-time curve (AUC[0-t]) of BAY1082439 after a single dose | Serial PK samples will be selected during cycle 1 day 1 (pre-dose and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, and 24 hours post-dose) and sparse samples during the rest of the cycle as well as in cycle 2

SECONDARY OUTCOMES:
Area under the concentration-time curve over the dosing interval (AUC[0-tau]) | PK parameters following single and repeat-dose administration in cycle 1
Maximum observed concentration (Cmax) | PK parameters following single and repeat-dose administration in cycle 1
Time of occurrence of Cmax (tmax) | PK parameters following single and repeat-dose administration in cycle 1
Terminal phase half-life (t1/2) | PK parameters following single and repeat-dose administration in cycle 1
Tumor response based on Response Evaluation Criteria in Solid Tumors, Version 1.1 | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Singapore, Singapore
- Seoul, South Korea
- Taipei, Taiwan